CLINICAL TRIAL: NCT00889356
Title: Phase III, Open Label, Randomized, Multicenter Study to Evaluate Efficacy, Tolerability & Safety of Combination of Clindamycin 100mg and Ketoconazole 400mg in Vaginal Capsules, Compared to Combination of Tetracycline 100mg and Amphotericin B 50mg in Vaginal Cream for the Treatment of Bacterial Vaginosis and Candidiasis Isolatedly or in Association (Mixed-Type Vaginosis)
Brief Title: Evaluate Efficacy, Tolerability & Safety of Combination of Clindamycin and Ketoconazole for the Treatment of Mixed-Type Vaginosis, Bacterial Vaginosis and Candidiasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zodiac Produtos Farmaceuticos S.A. (Industry)
Responsible Party: Julio Cesar Nophal de Carvalho, Zodiac Produtos Farmaceuticos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZD 002-08
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Candidiasis; Bacterial Vaginosis
MeSH Terms: conditions — Candidiasis; Vaginosis, Bacterial | interventions — Clindamycin; Ketoconazole; Tetracycline; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clindamycin 100mg and Ketoconazole 400mg (Experimental)
  Interventions: Drug: Clindamycin 100mg and Ketoconazole 400mg
- Tetracycline 100mg and Amphotericin B 50mg (Active Comparator)
  Interventions: Drug: Tetracycline 100mg and Amphotericin B 50mg

INTERVENTIONS:
Drug: Clindamycin 100mg and Ketoconazole 400mg — 1 vaginal capsule once a day at night
  Arms: Clindamycin 100mg and Ketoconazole 400mg
Drug: Tetracycline 100mg and Amphotericin B 50mg — One full applicator, once a day at night
  Arms: Tetracycline 100mg and Amphotericin B 50mg

SUMMARY:
The purpose of this study is to determine the Efficacy, Tolerability & Safety of Combination of Clindamycin 100mg and Ketoconazole 400mg in Vaginal Capsules, used for 7 consecutive days in patients with Mixed-Type Vaginosis compared to Combination of Tetracycline 100mg and Amphotericin B 50mg in Vaginal Cream.

ELIGIBILITY:
Inclusion Criteria:

* Mixed-type vaginosis
* Bacterial vaginosis
* Candidiasis

Exclusion Criteria:

* Pregnancy
* Vaginal bleeding
* History of recurrent vaginosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy based on cure rate evaluated by clinical and laboratory criteria. | 7 days

SECONDARY OUTCOMES:
Tolerability based on adverse events reports and patient's information | 7 days
Safety based on adverse events reports and laboratory criterion | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Bonassi Machado, MD, Principal Investigator — CRM Regional Council of Medicine
Locations (1):
- Vox Femina, Jundiaí, São Paulo, Brazil